CLINICAL TRIAL: NCT02334995
Title: The Biofeedback Therapy in Solitery Rectal Ulser Patients
Brief Title: The Biofeedback Therapy in Solitery Rectal Ulser Patients BIOFEEDBACK THERAPY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Serhat Bor, Professor Dr, Ege University
Other Study IDs: SRUS-BF; SRUS-BF (Registry Identifier: SRUS-BF)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Rectal Ulcer
Keywords: solitery rectal ulcer; biofeedback; dissynergy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dissynergic defecation causes solitery rectal ulcer. The biofeedback therapy improves dissynegy and heals soliter rectal ulcer.

DETAILED DESCRIPTION:
dyssynergia treating ulcers caused by treatment with biofeedback

ELIGIBILITY:
Inclusion Criteria:

* solitary rectal ulcer in rectosigmoidoscopy
* type 1 or 3 dissynergic defecation
* to accept to participate to study and sign informed consent

Exclusion Criteria:

* previously applied biofeedback
* serious psychiatric disorder
* previous anorectal surgery
* the presence of active malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solitary rectal ulser
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
ulcer diameter shrinkage | 6-8 weeks
  ulcer diameter measured in rectosigmoidoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Bor, Principal Investigator
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)